CLINICAL TRIAL: NCT03120390
Title: Reducing Metabolic Dysregulation in Obese Latina Breast Cancer Survivors Using Physical Activity: The ROSA Trial (Phase II, Randomized Controlled Trial for Early Stage Breast Cancer Survivors)
Brief Title: Physical Activity in Reducing Metabolic Dysregulation (MetD) in Obese Latina Breast Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1B-15-6; NCI-2017-00532 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-15-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-04-13; First posted 2017-04-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Cancer Survivor; Central Obesity; No Evidence of Disease
MeSH Terms: conditions — Obesity, Abdominal | interventions — Practice Guidelines as Topic; Standard of Care; Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Group I (PCT) (Experimental): Patients undergo supervised exercise sessions comprising of AE over 30 minutes and RE over 25 minutes 3 days per week for 24 weeks. Patients are encouraged to complete AE at home over 20 minutes 1 day per week. Patients receive a Polar heart rate monitor to monitor heart rate during the AE sessions.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Device: Monitoring Device; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (PAT) (Experimental): Patients undergo supervised exercise sessions comprising of AE over 45-60 minutes 3 days per week for 24 weeks. Patients are encouraged to complete AE at home over 20 minutes 1 day per week. Patients receive a Polar heart rate monitor to monitor heart rate during the AE sessions.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Device: Monitoring Device; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group III (usual care) (Active Comparator): Patients undergo usual care. Beginning 24 weeks, patients may undergo supervised exercise sessions comprising of AE and RE as in Group I.
  Interventions: Other: Best Practice; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Undergo usual care
  Other Names: standard of care; standard therapy
  Arms: Group III (usual care)
Behavioral: Exercise Intervention — Undergo AE
  Arms: Group I (PCT); Group II (PAT)
Behavioral: Exercise Intervention — Undergo RE
  Arms: Group I (PCT)
Other: Laboratory Biomarker Analysis — Correlative studies
Device: Monitoring Device — Receive Polar heart rate monitor
  Other Names: Monitor
  Arms: Group I (PCT); Group II (PAT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well physical activity works in reducing metabolic dysregulation in obese Latina breast cancer survivors. Physical activity may improve fitness and lessen metabolic disease (such as coronary artery disease, stroke, and type 2 diabetes) risk factors in patients who have breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effects of a 6-month progressive combined training (PCT) program on metabolic dysregulation (MetD) in centrally obese latina breast cancer survivors (LBCS).

SECONDARY OBJECTIVES:

I. To determine whether improved physical fitness and health-related measures from a 6-month PCT program are associated with reductions in MetD in centrally obese LBCS.

II. To determine whether MetD status and physical fitness can be maintained following a 6-month follow-up period and to establish predictors of exercise behavior in LBCS.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I (PROGRESSIVE COMBINED TRAINING [PCT]): Patients undergo supervised exercise sessions comprising of aerobic exercise (AE) over 30 minutes and resistance exercise (RE) over 25 minutes 3 days per week for 24 weeks. Patients are encouraged to complete AE at home over 20 minutes 1 day per week. Patients receive a Polar heart rate monitor to monitor heart rate during the AE sessions.

GROUP II (PROGRESSIVE AEROBIC TRAINING [PAT]): Patients undergo supervised exercise sessions comprising of AE over 45-60 minutes 3 days per week for 24 weeks. Patients are encouraged to complete AE at home over 20 minutes 1 day per week. Patients receive a Polar heart rate monitor to monitor heart rate during the AE sessions.

GROUP III (USUAL CARE): Patients undergo usual care. Beginning 24 weeks, patients may undergo supervised exercise sessions comprising of AE and RE as in Group I.

After completion of study, patients are followed up at 37 and 49 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (stage I-III) breast cancer
* Self-identify as Latina
* Have undergone a lumpectomy or mastectomy
* Have received and completed neoadjuvant or adjuvant cytotoxic chemotherapy and/or radiation therapy within the past 12 months
* Have no evidence of cancer disease after treatment (confirmed by their treating physician)
* Able to initiate a supervised exercise program (free from any cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity; obtains clearance from physician to confirm status)
* Are centrally obese with the following criteria (determined by study team at eligibility screening): body mass index (BMI) > 30 kg/m^2 (calculated using height and weight) or body fat > 30% (estimated by bioelectrical impedance), and waist circumference > 35 inches (in)
* Free from history of chronic disease including severe diabetes (glycosylated hemoglobin [HgA1c] > 7% requiring a pharmacologic intervention), uncontrolled hypertension or thyroid disease (obtains clearance from physician to confirm status)
* Have not experienced a weight reduction >= 10% within past 6 months; and body weight has remained stable for the past 4 weeks
* Currently participate in less than 60 minutes of physical activity/week
* No planned reconstructive surgery with flap repair during trial and follow-up period
* May use adjuvant endocrine therapy if use will be continued for duration of study period
* Does not smoke (no smoking during previous 12 months)
* Willing to travel to the exercise facility at University of Southern California (USC) (parking fees and public transportation permits will be provided)

Exclusion Criteria:

* Currently pregnant
* History of chronic disease including uncontrolled diabetes, uncontrolled hypertension or uncontrolled thyroid disease; women using metformin to manage diabetes will be excluded from the trial
* Weight reduction >= 10% within past 6 months
* Metastatic disease
* Planned reconstructive surgery with flap repair during trial and follow-up period
* Cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change in MetD | From week 25 to week 49
  Insulin resistance (IR) measured by Homeostasis Model Assessment (HOMA) will be assessed from baseline.

SECONDARY OUTCOMES:
Change in cardiorespiratory fitness | Baseline to week 49
  Subjects will be instructed to walk comfortably (so they are able to talk while walking) on a treadmill for 4 minutes and heart rate will be measured at the end of the test to estimate maximal oxygen uptake.
Change in functional capacity | Baseline to week 49
  1). Hand grip strength: Grip strength will be measured using a hand-held dynamometer on the participant's dominant hand. The subject will be asked to grip the handle of the dynamometer with one hand using as much grip pressure as possible while holding for 2 seconds; 2). Y Balance Test: All subjects will be required to complete the Y Balance by standing on a single limb and reach as far as possible with the opposite limb; 3). Modified Margaria-Kalamen Step Test will be used to test leg muscle power. Subjects will climb a flight of 10 stairs as quickly as possible, without missing a stair and will be evaluated based on time-to-completion and accuracy of completing all steps, given a total of 3 chances to complete the test as quickly as possible.
Change in muscle strength | Baseline to week 49
  The 10-repetition maximum (10-RM) method will test maximal voluntary strength for the following exercises: chest press, seated row, knee extension, knee flexion will be used to calculate maximum strength values for the resistance exercise intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, Ph.D., Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States